CLINICAL TRIAL: NCT04286191
Title: Characterization of Physiological Changes Induced Through Motor-evoked Potential Conditioning in People With Spinal Cord Injury
Brief Title: Physiological Changes Induced Through MEP Conditioning in People With SCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Aiko Thompson, Associate Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 00091457; 1R01NS114279-01 (NIH)
Record Dates: First submitted 2020-02-24; First posted 2020-02-26 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Spinal Cord Injuries; Neurological Injury; Paralysis; Spasticity, Muscle
Keywords: Corticospinal Tract; Neuroplasticity
MeSH Terms: conditions — Spinal Cord Injuries; Trauma, Nervous System; Paralysis; Muscle Spasticity | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Up-conditioning (UC) Group (Experimental)
  Interventions: Combination Product: Operant Conditioning
- Control (NC) Group (Sham Comparator)
  Interventions: Combination Product: Control Group

INTERVENTIONS:
Combination Product: Operant Conditioning — This is a training intervention in which the brain-spinal cord-muscle pathways are strengthened in individuals with incomplete spinal cord injury. Transcranial magnetic stimulation (TMS), a type of brain stimulation, will be used to elicit a muscle response from the tibialis anterior (TA), the muscle that lifts your toes and foot.
  Arms: Up-conditioning (UC) Group
Combination Product: Control Group — This is the control intervention, or the non-conditioning group. Transcranial magnetic stimulation (TMS), a type of brain stimulation, will be used to elicit a muscle response from the tibialis anterior (TA), the muscle that lifts your toes and foot.
  Arms: Control (NC) Group

SUMMARY:
The study team is currently recruiting volunteers who are interested in participating in a brain-spinal cord-muscle response training study that aims to better understand the changes that take place in the nervous system as a result of this type of training. After spinal cord injury, brain-to-muscle connections are often interrupted. Because these connections are important in movement control, when they are not working well, movements may be disturbed. Researchers have found that people can learn to strengthen these connections through training. Strengthening these connections may be able to improve movement control and recovery after injuries.

Research participants will be asked to stand, sit, and walk during the study sessions. Electrodes are placed on the skin over leg muscles for monitoring muscle activity. For examining brain-to-muscle connections, the study team will use transcranial magnetic stimulation. The stimulation is applied over the head and will indirectly stimulate brain cells with little or no discomfort.

Participation in this study requires approximately three sessions per week for four months, followed by two to three sessions over another three months. Each session lasts approximately 1 hour.

ELIGIBILITY:
Inclusion Criteria:

* Neurologically stable (>1 year post SCI)
* Medical clearance to participate
* Ability to ambulate at least 10 m with or without an assistive device (except for parallel bars)
* Signs of weak ankle dorsiflexion at least unilaterally
* Expectation that current medication will be maintained without change for at least 3 months; stable use of anti-spasticity medication is accepted

Exclusion Criteria:

* motoneuron injury
* known cardiac condition (e.g., history of myocardial infarction, congestive heart failure, pacemaker use)
* medically unstable condition
* cognitive impairment
* history of epileptic seizures
* metal implants in the cranium
* implanted biomedical device in or above the ches (e.g., a cardiac pacemaker, cochlear implant)
* no measurable MEP elicited
* unable to produce any voluntary TA EMG activity
* extensive use of functional electrical stimulation to the leg on a daily basis
* pregnancy (due to changes in weight and posture and potential medical instability)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Change in the excitability/strength of the brain-spinal cord-muscle pathway at the brain level as measured by the MEP recruitment curve--Studied Leg | Baseline through 3 months post intervention
  An increased maximum MEP size (mV) would indicate increased excitability/strength of the brain-spinal cord-muscle pathway
Change in the cortical map of the Tibialis Anterior: identifying the size (cm2) of the area of the brain that controls the tibialis anterior, the muscle that raises the toes and foot--Studied Leg | Baseline through 3 months post intervention
  Reorganization of the TA cortical map would suggest that operant conditioning of the muscle response changes the brain. Knowing if and how the brain changes will help investigators understand the potential impact of this type of training.
Change in the excitability/strength of the brain-spinal cord-muscle pathway at the spinal-cord level as measured by the Cervicomedullary MEP (CMEP) size--Studied Leg | Baseline through 3 months post intervention
  An increase in the size of the CMEP (mV) elicited at a fixed stimulus intensity would indicate increased excitability/strength at the spinal cord level
Change in excitability of the excitability of the brain as measured by Short Interval Intra-cortical Inhibition (SICI) | Baseline through 3 months post intervention
  Decreased SICI indicates increased excitability in the brain
Change in reflex activity as measured by the H-reflex amplitude (mV) in response to nerve stimulation--Studied Leg | Baseline through 3 months post intervention
  Decreased H-reflex amplitude indicates reduced reflex activity and a more normal reflex response to muscle activity
Change in excitability/strength of the spinal cord-muscle pathway as measured by Change in F-wave amplitude (mV) and F-wave occurrence (out of 30 trials) in response to nerve stimulation--Studied Leg | Baseline through 3 months post intervention
  Increased F-wave amplitude and/or occurrence indicates increased excitability/strength of the spinal cord-muscle pathway
Change in the ability to activate the muscle that lifts the toes during the swing-phase of walking as measured by tibialis anterior EMG amplitude (mv)--Studied Leg | Baseline through 3 months post intervention
  Increased EMG amplitude indicates greater activation of the muscle, which could indicate an increased ability to lift the toes during the swing-phase of walking
Change in ankle joint motion during walking (deg)--Studied Leg | Baseline through 3 months post intervention
  Ankle range of motion over the step cycle (in deg); Ankle peak flexion angle (in deg); Ankle angle at foot contact (in deg); Median ankle angle over the step cycle (in deg)
Change in walking speed (m/s) as measured by the 10-meter walk test | Baseline through 3 months post intervention
  Speed of the participant's fastest comfortable walking speed across 10 meters. Decreased time (sec) demonstrates increased walking speed (m/s)
Change in walking distance (meters) as measured by the 6-minute walk test | Baseline through 3 months post intervention
  The distance walked in 6 minutes in measured. The participant is asked to walk at his/her fastest comfortable speed on an indoor walkway.

SECONDARY OUTCOMES:
Change in the excitability/strength of the brain-spinal cord-muscle pathway at the brain level as measured by the MEP recruitment curve--Contralateral Leg | Baseline through 3 months post intervention
  An increased maximum MEP size (mV) would indicate increased excitability/strength of the brain-spinal cord-muscle pathway
Change in the cortical map of the Tibialis Anterior: identifying the size (cm2) of the area of the brain that controls the tibialis anterior, the muscle that raises the toes and foot--Contralateral Leg | Baseline through 3 months post intervention
  Reorganization of the TA cortical map would suggest that operant conditioning of the muscle response changes the brain. Knowing if and how the brain changes will help investigators understand the potential impact of this type of training.
Change in the excitability/strength of the brain-spinal cord-muscle pathway at the spinal-cord level as measured by the Cervicomedullary MEP (CMEP) size--Contralateral Leg | Baseline through 3 months post intervention
  An increase in the size of the CMEP (mV) elicited at a fixed stimulus intensity would indicate increased excitability/strength at the spinal cord level
Change in reflex activity as measured by the H-reflex amplitude (mV) in response to nerve stimulation--Contralateral Leg | Baseline through 3 months post intervention
  Decreased H-reflex amplitude indicates reduced reflex activity and a more normal reflex response to muscle activity
Change in excitability/strength of the spinal cord-muscle pathway as measured by Change in F-wave amplitude (mV) and F-wave occurrence (out of 30 trials) in response to nerve stimulation--Contralateral Leg | Baseline through 3 months post intervention
  Increased F-wave amplitude and/or occurrence indicates increased excitability/strength of the spinal cord-muscle pathway
Change in the ability to activate the muscle that lifts the toes during the swing-phase of walking as measured by tibialis anterior EMG amplitude (mv)--Contralateral Leg | Baseline through 3 months post intervention
  Increased EMG amplitude indicates greater activation of the muscle, which could indicate an increased ability to lift the toes during the swing-phase of walking
Change in ankle joint motion during walking (deg)--Studied Leg | Baseline through 3 months post intervention
  Ankle range of motion over the step cycle (in deg); Ankle peak flexion angle (in deg); Ankle angle at foot contact (in deg); Median ankle angle over the step cycle (in deg)
Change in knee joint motion during walking (deg)--Both Legs | Baseline through 3 months post intervention
  Knee range of motion over the step cycle (in deg); knee peak flexion angle (in deg); knee peak extension angle (in deg); knee angle at foot contact (in deg); median knee angle over the step cycle (in deg)
Change in hip joint motion during walking (deg)--Both Legs | Baseline through 3 months post intervention
  Hip range of motion over the step cycle (in deg); hip peak flexion angle (in deg); hip peak extension angle (in deg); hip angle at foot contact (in deg); median hip angle over the step cycle (in deg)
Changes in reflexes and muscle activation during walking as measured by H-reflex size and cutaneous reflex size | Baseline through 3 months post intervention
  Decreased H-reflex response and decreased radiating threshold of the cutaneous reflex would reflect reflex activity that is more similar to individuals without neurological injury

CONTACTS AND LOCATIONS:
Overall Officials: Aiko K Thompson, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-03-28): https://cdn.clinicaltrials.gov/large-docs/91/NCT04286191/ICF_000.pdf